CLINICAL TRIAL: NCT04823533
Title: A Psychophysiological Study of the Bidirectional Communication Mechanisms Between the Brain and the Gastrointestinal System and Its Effects on Well-being
Brief Title: Improving Wellbeing Through the Brain-Gut-Microbiota Axis
Acronym: IBMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: University of Chile (Other); Instituto de Nutrición y Tecnología de los Alimentos (Other); University Diego Portales (Other); Lallemand SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 181014002
Record Dates: First submitted 2021-03-05; First posted 2021-03-30 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Healthy Lifestyle
Keywords: Microbiota; Brain-gut; Wellbeing; Interoception; Probiotic; Electrophysiology

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): A probiotic formulation containing two well-documented probiotic strains. The finished product is a lyophilized powder packaged in single-dose sticks sachets Excipients used were as follows: xylitol, maltodextrin, plum flavor, and malic acid.
  Interventions: Dietary Supplement: Probiotic-placebo supplement
- Placebo (Placebo Comparator): Placebo formulation containing only the excipients used were as follows: xylitol, maltodextrin, plum flavor, and malic acid.
  Interventions: Dietary Supplement: Probiotic-placebo supplement

INTERVENTIONS:
Dietary Supplement: Probiotic-placebo supplement — A probiotic formulation containing two well-documented probiotic strains. The finished product is a lyophilized powder packaged in single-dose sticks sachets Excipients used were as follows: xylitol, maltodextrin, plum flavor, and malic acid.

SUMMARY:
Well-being is a state defined as the optimal psychological functioning and the experience associated with it, integrating physical and subjective factors. It has been suggested that the bidirectional interaction between the brain and the rest of the body is fundamental in the regulation of wellbeing levels. In particular, the gastrointestinal system (modulated by the microbiota) sends information that is integrated by the brain, affecting its functioning and mental processes. However, the mechanism of such communication is still unknown. The aim of this proposal is to study the different ways in which psychological processes can influence gut signals and vice versa, and how this relationship might be trained or modified in order to improve wellbeing.

DETAILED DESCRIPTION:
Within the field of Psychology and Contemplative Sciences, the relationship and interdependence between the brain and body have been one of the most prevalent questions when it comes to understanding the psychobiological mechanisms underlying human behavior. It is proposed that the brain should be seen as a dynamic, complex, and self-organized system, which is closely coupled and integrated with whole-body signals, establishing a two-way communication axis. This has been evidenced through an increase in scientific research adopting an embodied perspective that considers both diverse brain measurements as well as signals from other parts of the body, such as the heart and the gastrointestinal system. Recent pieces of evidence have furthermore begun to reveal the different ways in which psychological processes can influence the body, and how this could be trained in order to improve wellness.

Interoception is a cognitive process developed to monitor the internal state of the body and it involves the continuous and dynamic integration of information from different (internal) origins, including respiratory, cardiac, and gastrointestinal systems. New research agendas have started to link interoception to wellbeing, and with the psychopathology of psychiatric conditions, from depression and autism to eating disorders. Interestingly, it has been shown that this ability can be trained through contemplative practices designed to improve body awareness, socio-affective and socio-cognitive capacity. Moreover, some interoceptive dimensions like thirst interoception might be affected by lifestyle and habits such as diet. Altogether, this evidence suggests that understanding the mechanism of brain-body integration represents a promising alternative to improve wellbeing and mental health.

One example of psychophysical integration that has taken much importance in recent years, due to its implications on wellbeing and mental health, is the one established between the brain and the gastrointestinal system. In particular, gut-microbiota research is acquiring special importance because of its implications in psychological states such as stress and anxiety, and psychiatric conditions like depression and autism. It has been shown that microbiota affects brain functioning through different pathways including neural, humoral, and endocrine. However, the mechanism of brain-gut-microbiota integration and its relationship to wellbeing is still unknown. The integration of information through large-scale oscillation coupling has been one of the most validated proposals regarding signal processing and communication. An oscillatory coupling between the brain and the gastrointestinal system was recently described, shedding light on a possible mechanism via which the gastrointestinal system constantly and instantaneously sends information to the brain, which in turn integrates this information either consciously or unconsciously, thus affecting mental processes.

This research proposal aims to study how the brain integrates information from the gut (regulated by the microbiota) and the relevance of this coupling on wellbeing. To do this, the oscillatory coupling between the electroencephalogram (EEG) and electrogastrogram (EGG) signals will be recorded and evaluated. EEGs and EGGs will be recorded under different interventions including training designed to increase interoceptive gastric awareness and treatment with probiotics to modify some microorganisms that have already been associated with mental health. The oscillatory coupling will be compared to the well-being observed after each of the interventions. In this investigation, wellbeing will be defined as optimal psychological functioning, integrating physical and subjective factors, and will be evaluated through different self-reported questionnaires.

Interventions related to improving body awareness and contemplative practices, in general, are helping to improve the levels of wellness around the world and in Chile, representing an accessible and cheap way to manage psychological conditions regardless of socioeconomic and demographic aspects, contributing to the development of new therapeutic strategies. Additionally, a strong relationship between diet, microbiota, and health has now been demonstrated. Thus, understanding the mechanism via which the microbiota communicates with the brain, the susceptibility of this communication to microbiota changes, and the relationship of this process with participants' diet could provide relevant information when making decisions related to eating habits and lifestyles.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults of ≥ 18 to & 65 years old of age.
2. Able to provide written consent.
3. Willing to provide stool samples and complete questionnaires, records, and diaries associated with the study
4. Willingness to discontinue consumption of probiotic supplements for the duration of the study.

Exclusion Criteria:

1. Concurrent consumption of probiotics. Subjects will be eligible for participation, however, after a four (4) week wash-out period.
2. Known to be pregnant or breastfeeding or planning on becoming pregnant in the next two (2) months.

   Positive pregnancy test in women of childbearing potential.
3. Use of antibiotic drugs (e.g., neomycin, rifaximin) within 1 month of the screening visit. The screened participant would be eligible to participate four (4) weeks after completing their course of antibiotics (wash-out period).
4. Subject with diabetes or metabolic diseases.
5. Subject with depression or psychiatric and neurological diseases.
6. Subject with IBS or gastrointestinal diseases.
7. Subject with immune disorders or with possible immune-deficient status (e.g. due to surgery).
8. Milk or soy allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) at baseline | Week 0
  The subjective experience associated with emotional regulation will be measured. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure).
Difficulties in Emotion Regulation Scale (DERS) after intervention | Week 4
  The subjective experience associated with emotional regulation will be measured. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post)
Difficulties in Emotion Regulation Scale (DERS) - follow up | Week 12
  The subjective experience associated with emotional regulation will be measured. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
Ryff Scales of Psychological Well-Being (PWB) at baseline | Week 0
  The scale measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure)
Ryff Scales of Psychological Well-Being (PWB) post intervention | Week 4
  The scale measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post)
Ryff Scales of Psychological Well-Being (PWB) - follow-up | Week 12
  The scale measures six aspects of wellbeing and happiness: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
Satisfaction With Life Scale (SWLS) at baseline | Week 0
  The Satisfaction With Life Scale (SWLS) was developed to assess satisfaction with the respondent's life as a whole. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure).
Satisfaction With Life Scale (SWLS) post intervention | Week 4
  The Satisfaction With Life Scale (SWLS) was developed to assess satisfaction with the respondent's life as a whole. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post)
Satisfaction With Life Scale (SWLS) - follow-up | Week 12
  The Satisfaction With Life Scale (SWLS) was developed to assess satisfaction with the respondent's life as a whole. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
The State-Trait Anxiety Inventory (STAI) - State at baseline | Week 0
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. For this experiment, the anxiety assessment will be restricted exclusively to the state. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure).
The State-Trait Anxiety Inventory (STAI) - State post intervention | Week 4
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. For this experiment, the anxiety assessment will be restricted exclusively to the state. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post)
The State-Trait Anxiety Inventory (STAI) - State - follow-up | Week 12
  The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. For this experiment, the anxiety assessment will be restricted exclusively to the state. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
Positive and Negative Affect Schedule (PANAS) at baseline | Week 0
  The Positive and Negative Affect Schedule (PANAS) comprises two mood scales, one that measures positive affect and the other which measures negative affect. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure).
Positive and Negative Affect Schedule (PANAS) post intervention | Week 4
  The Positive and Negative Affect Schedule (PANAS) comprises two mood scales, one that measures positive affect and the other which measures negative affect. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post).
Positive and Negative Affect Schedule (PANAS) - follow-up | Week 12
  The Positive and Negative Affect Schedule (PANAS) comprises two mood scales, one that measures positive affect and the other which measures negative affect. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
The Five Facet Mindfulness Questionnaire (FFMQ) at baseline | Week 0
  The Five Facet Mindfulness Questionnaire is an established and valid psychometric self-assessment for mindfulness. The five facets are: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure).
The Five Facet Mindfulness Questionnaire (FFMQ) post intervention | Week 4
  The Five Facet Mindfulness Questionnaire is an established and valid psychometric self-assessment for mindfulness. The five facets are: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post).
The Five Facet Mindfulness Questionnaire (FFMQ) - follow-up | Week 12
  The Five Facet Mindfulness Questionnaire is an established and valid psychometric self-assessment for mindfulness. The five facets are: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
Gut microbiota | Week 0
  Plastic containers with the stool sample will be stored at -20 ° C in a refrigerator for the maintenance of biological samples located in the EPUC. Genomic DNA will be extracted from each sample and amplified in two steps. In the first step, a particular region encoding for a part of the 16s ribosomal RNA typical of prokaryotic organisms will be amplified by PCR. In a second step, a second PCR will be carried out in order to add the primers required for future sequencing. Finally, the results of the amplification will be quantified using qPCR, and will be stored in genomic libraries for subsequent sequencing and bioinformatic analysis [50]. This procedure will be performed to obtain the total bacterial colonies present in the faecal samples.
Water load test (Gastric Interoception) at baseline | Week 0
  Briefly, participants will have to drink room-temperature water for a period of 5 minutes until they feel signs of satiation at the beginning and then until feeling completely full of water. Different interoceptive indicators can be obtained using the water volumes required for feeling satiated and full.
  Participants will be evaluated by performing the task at baseline
Water load test (Gastric Interoception) post intervention | Week 4
  Briefly, participants will have to drink room-temperature water for a period of 5 minutes until they feel signs of satiation at the beginning and then until feeling completely full of water. Different interoceptive indicators can be obtained using the water volumes required for feeling satiated and full.
  Participants will be evaluated by performing the task after 4 weeks of intervention
Water load test (Gastric Interoception) - follow-up | Week 12
  Briefly, participants will have to drink room-temperature water for a period of 5 minutes until they feel signs of satiation at the beginning and then until feeling completely full of water. Different interoceptive indicators can be obtained using the water volumes required for feeling satiated and full.
  Participants will be evaluated by performing the task after 12 weeks since the baseline measure (follow-up)
Multidimensional questionnaire of interoceptive awareness (MAIA) at baseline | Week 0
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception by self-report. These are labeled Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trust
  For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire at the beginning of the experiment (baseline measure)
Multidimensional questionnaire of interoceptive awareness (MAIA) post intervention | Week 4
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception by self-report. These are labeled Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trust
  For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 4 weeks of the intervention (Post)
Multidimensional questionnaire of interoceptive awareness (MAIA) follow-up | Week 12
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is an 8-scale state-trait questionnaire with 32 items to measure multiple dimensions of interoception by self-report. These are labeled Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trust
  For this, aspects of the subjective experience of the participants will be evaluated at the present time or in the daily life of their lives by completing the questionnaire after 12 weeks since the baseline measure (follow-up)
Brain-gut coupling using the modulation index | Week 0
  The brain-gut oscillatory coupling is one outcome that is obtained by measuring the power amplitude of the Electroencephalographic (EEG) and phase of the electrogastrographic (EGG) activity.
  The Brain-gut oscillatory coupling is obtained by calculating a modulation index between the phase of the EGG slow frequency gastric oscillations (0.05 Hz) and the power amplitude of EEG alpha oscillations (8-12 Hz). The modulation index is a measurement that indicates in which extend the phase of slow gastric oscillations modulate the amplitude of alpha waves For the EEG activity, 64 active electrodes will be positioned on a cap located on the participant's head. For the EGG record, a set of 16 skin electrodes will be positioned on the abdomen as described in Richter, Babo-Rebelo.

CONTACTS AND LOCATIONS:
Locations (1):
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile